CLINICAL TRIAL: NCT00435045
Title: A Randomized, Double-Blind, Placebo-Controlled, Forced Titration Study to Assess the Efficacy and Safety of Omacor, Co-Administered With Open-Label Atorvastatin Therapy, in Hypertriglyceridemic Subjects
Brief Title: Evaluation of Efficacy and Safety of Omacor, Co-Administered With Atorvastatin, in Subjects With Hypertriglyceridemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OM9L
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Results first posted 2009-05-12 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Hypertriglyceridemia
Keywords: Lovaza; Hyperlipidemias; Triglycerides; Lipids; omega-3 fatty acids; Hypercholesterolemia; Hypertriglyceridemia; omega-3-acid ethyl esters; Omacor; Dyslipidemias
MeSH Terms: conditions — Hypertriglyceridemia; Hyperlipidemias; Hypercholesterolemia; Dyslipidemias | interventions — Omacor; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- atorvastatin arm (Active Comparator): atorvastatin + placebo
  Interventions: Drug: atorvastatin
- Lovaza arm (Experimental): Lovaza + atorvastatin
  Interventions: Drug: Lovaza (omega-3-acid ethyl esters) [formerly known as Omacor] plus atorvastatin

INTERVENTIONS:
Drug: Lovaza (omega-3-acid ethyl esters) [formerly known as Omacor] plus atorvastatin — Lovaza + atorvastatin
  Arms: Lovaza arm
Drug: atorvastatin — atorvastatin + placebo
  Other Names: Lovaza (omega-3-acid ethyl esters) [formerly known as Omacor] plus atorvastatin
  Arms: atorvastatin arm

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Omacor (omega-3-acid ethyl esters) combined with atorvastatin for lowering non-high-density lipoprotein cholesterol (non-HDL-C) in hypertriglyceridemic subjects.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, parallel-group study design with eleven clinic visits (one screening visit, three lead-in/baseline visits, and seven treatment visits) After a 4-week diet only lead-in period, subjects with a triglyceride (TG) level in the high to very high range and with non-HDL-C level above NCEP ATPIII goals will be randomized to receive either open-label atorvastatin 10 mg per day plus double-blinded Lovaza 4g (4 x 1g capsules) per day OR open-label atorvastatin 10 mg per day plus a double-blinded matching placebo (4 corn oil capsules per day) for 8 weeks After the initial 8-week treatment period, the dose of open-label atorvastatin will be titrated to 20 mg per day (with the Lovaza or matching placebo corn oil doses remaining at 4 capsules per day) for an additional 4 weeks At Week 12, a second open-label titration to 40 mg of open-label atorvastatin per day will be maintained for an additional 4 weeks (again with the Lovaza or matching placebo corn oil doses remaining at 4 capsules per day)

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18-79 years, inclusive
* Fasting, untreated non-high-density lipoprotein cholesterol (non-HDL-C) level above NCEP ATPIII goals
* Fasting, untreated triglyceride (TG) level in the high to very high range
* Provide written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Pregnancy
* Use of lipid-altering drugs which cannot be stopped
* History of certain cardiovascular conditions or cardiac surgery within prior 6 months
* Body mass index above 40 kg per square meter
* Allergy or sensitivity to omega-3 fatty acids or to statin drugs
* Poorly-controlled conditions including diabetes, hypertension, or thyroid disease
* Certain muscle, liver, kidney, lung, or gastrointestinal conditions
* Certain medications
* Active cancers treated within prior 2 years (except non-melanoma skin cancer)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2007-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bays HE, McKenney J, Maki KC, Doyle RT, Carter RN, Stein E. Effects of prescription omega-3-acid ethyl esters on non--high-density lipoprotein cholesterol when coadministered with escalating doses of atorvastatin. Mayo Clin Proc. 2010 Feb;85(2):122-8. doi: 10.4065/mcp.2009.0397. PMID 20118387
- [Derived] Maki KC, Bays HE, Dicklin MR, Johnson SL, Shabbout M. Effects of prescription omega-3-acid ethyl esters, coadministered with atorvastatin, on circulating levels of lipoprotein particles, apolipoprotein CIII, and lipoprotein-associated phospholipase A2 mass in men and women with mixed dyslipidemia. J Clin Lipidol. 2011 Nov-Dec;5(6):483-92. doi: 10.1016/j.jacl.2011.09.001. Epub 2011 Sep 13. PMID 22108152
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: OM9L — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: OM9L — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: OM9L — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: OM9L — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: OM9L — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: OM9L — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: OM9L — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Lovaza(Omacor) + Atorvastatin: Subjects who met all study requirements after screening visit and who were randomized to receive 4 gms Lovaza (Omega-3-acid ethyl esters) + Atorvastatin 10 mgs for 8 weeks, then 4 gms Lovaza + Atorvastatin 20 mgs for 4 weeks, then 4 gms Lovaza + Atorvastatin 40 mgs for 4 additional weeks.
- Placebo + Atorvastatin: Subjects who met all study requirements after screening visit and who were randomized to receive Placebo + Atorvastatin 10 mgs for 8 weeks, then Placebo + Atorvastatin 20 mgs for 4 weeks, then Placebo + Atorvastatin 40 mgs for 4 additional weeks.
Period: Weeks 1-8 / 10 mg Dose Level
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Started | 123 | 122
Completed | 118 | 118
Not Completed | 5 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Family Crisis - could not participate | 1 | 0
Not completed — Requirement for Excluded Medications | 0 | 1
Period: Weeks 9-12 / 20mg Dose Level
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Started | 118 | 118
Completed | 113 | 113
Not Completed | 5 | 5
Not completed — Adverse Event | 4 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Weeks 13-16 / 40mg Dose Level
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Started | 113 | 113
Completed | 108 | 111
Not Completed | 5 | 2
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Per Sponsors Request | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin | Total
Number analyzed (Participants) | 123 | 122 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (9.64) | 56.0 (10.84) | 56.1 (10.23)
Gender [Count of Participants; unit: Participants]
  Female | 52 | 51 | 103
  Male | 71 | 71 | 142
Race/Ethnicity, Customized [Number; unit: participants]
  White | 108 | 110 | 218
  Black or African American | 6 | 4 | 10
  Asian | 8 | 4 | 12
  American Indian or Alaskan Native | 0 | 1 | 1
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Non-white | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Non-high density lipoprotein cholesterol is the Total Cholesterol minus the HDL(high density lipoproteins or the sum of the LDL, VLDL and IDL. That is, Low Density Lipoproteins, Very Low Density Lipoproteins and Intermediate Density Lipoproteins.
Time Frame: Baseline and Week 8
Population: Modified Intent To Treat (MITT) Population - all randomized subjects who took at least 1 dose of study medication and provided at least 1 post-randomization efficacy data point. Only subjects with non-missing baseline and endpoint values are included.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 122 | 121
percent change | -40.2 [-45.3 to -32.5] | -33.7 [-39.6 to -28.3]
Statistical Analysis 1: Comparison: Lovaza(Omacor) + Atorvastatin vs Placebo + Atorvastatin; Test type: Non-Inferiority or Equivalence — Non-inferiority of the non-HDL-C response was assessed by calculating the 2-sided 90% and 95% confidence intervals (CIs)for each difference in response based on comparing the effects of increases in atorvastatin dose on the percent changes from baseline to the end of each atorvastatin period, a repeated-ANOVA model was used; p = 0.0002, ANOVA

2. Secondary Outcome: Percent Change in Total Cholesterol (TC) From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Total Cholesterol is the sum of the High Density Lipoproteins (HDL), Low Density Lipoproteins (LDL), Very Low Density Lipoproteins (VLDL), and Intermediate Density Lipoproteins (IDL).
Time Frame: Baseline and Week 8
Population: Modified Intent To Treat Population - all randomized subjects who took at least 1 dose of study medication and provided at least 1 post-randomization efficacy data point. Only subjects with non-missing baseline and endpoint values are included.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 122 | 121
percent change | -31.5 [-36.0 to -25.3] | -27.4 [-31.7 to -22.2]

3. Secondary Outcome: Percent Change in High Density Lipoprotein (HDL)Cholesterol From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: HDL - A complex of lipids and proteins in approximately equal amounts that functions as a transporter of cholesterol in the blood. High levels are associated with a decreased risk of atherosclerosis and coronary heart disease.
  High density lipoprotein cholesterol is the Total Cholesterol minus the sum of the LDL, VLDL and IDL.
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 122 | 121
percent change | 12.4 [3.6 to 22.9] | 10.0 [-1.2 to 16.3]

4. Secondary Outcome: Percent Change in Low Density Lipoprotein (LDL) Cholesterol (Beta-quantification) From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: LDL - A complex of lipids and proteins, with greater amounts of lipid than protein, that transports cholesterol in the blood. High levels are associated with an increased risk of atherosclerosis and coronary heart disease.
Time Frame: Baseline and Week 8
Population: Modified Intent To Treat Population - all randomized subjects who took at least 1 dose of study medication and provided at least 1 post-randomization efficacy data point. Please note: processing errors, inadequate sample volume, sample and shipment storage issues etc., resulted in some MITT subjects without data.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 122 | 120
percent change | -29.3 [-41.1 to -18.4] | -31.5 [-41.4 to -23.4]

5. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Triglycerides - A naturally occurring ester of three fatty acids and glycerol that is the chief constituent of fats and oils.
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 122 | 121
percent change | -45.4 [-55.3 to -34.9] | -26.9 [-38.7 to -14.4]

6. Secondary Outcome: Percent Change in Very Low Density Lipoproteins (VLDL) Cholesterol From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: VLDL - very-low-density lipoprotein: a plasma lipoprotein with a high lipid content, associated with atherosclerosis.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 122 | 120
percent change | -54.3 [-66.7 to -36.7] | -37.0 [-50.9 to -17.8]

7. Secondary Outcome: Percent Change in Apolipoprotein-A-1 From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Apolipoprotein A1 - major protein component of high density lipoprotein (HDL) in plasma. The protein promotes cholesterol efflux from tissues to the liver for excretion.
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 122 | 121
percent change | -0.3 [-7.0 to 9.0] | 1.5 [-4.5 to 10.4]

8. Post Hoc Outcome: Percent Change in Apolipoprotein-B From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Apolipoprotein B is the primary apolipoprotein of low density lipoproteins (LDL or "bad cholesterol"), which is responsible for carrying cholesterol to tissues.
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 122 | 121
percent change | -32.1 [-40.1 to -24.2] | -30.7 [-36.0 to -23.0]

9. Secondary Outcome: Percent Change in Apolipoprotein C-III From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Apolipoprotein C-III (APOC3) is a very low density lipoprotein (VLDL) protein. APOC3 inhibits lipoprotein lipase and hepatic lipase; it is thought to delay catabolism of triglyceride-rich particles.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 119 | 119
percent change | -29.4 [-36.8 to -17.4] | -16.0 [-27.3 to 0.0]

10. Secondary Outcome: Percent Change in Total Cholesterol/High Density Lipoprotein Cholesterol Ratio From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Total cholesterol/High density lipoprotein cholesterol
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 122 | 121
percent change | -38.3 [-44.9 to -31.9] | -34.5 [-40.3 to -25.0]

11. Secondary Outcome: Percent Change in Triglycerides/High Density Lipoprotein Cholesterol Ratio From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 122 | 121
percent change | -51.9 [-62.4 to -39.8] | -34.0 [-47.3 to -14.9]

12. Secondary Outcome: Percent Change in Docosahexaenoic Acid (DHA) From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Docosahexaenoic Acid is an omega-3 essential fatty acid.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 101 | 103
percent change | 85.5 [49.4 to 125.6] | 4.2 [-5.7 to 13.4]

13. Secondary Outcome: Percent Change in Eicosapentaenoic Acid (EPA) From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Eicosapentaenoic acid (EPA) is one of several omega-3 fatty acids used by the body. It is found in cold water fatty fish and in fish oil supplements, along with docosahexaenoic acid (DHA). Omega-3 fatty acids are part of a healthy diet that helps lower risk of heart disease.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 101 | 103
percent change | 402.2 [276.8 to 570.8] | -5.6 [-20.0 to 14.9]

14. Secondary Outcome: Percent Change in Low Density Lipoprotein Particle Concentration Total From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Low-density lipoproteins - A complex of lipids and proteins, with greater amounts of lipid than protein, that transports cholesterol in the blood. High levels are associated with an increased risk of atherosclerosis and coronary heart disease.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 119 | 118
percent change | -34.6 [-42.9 to -24.0] | -32.2 [-41.2 to -23.5]

15. Secondary Outcome: Percent Change in Low Density Lipoprotein Particle Size From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Low-density lipoproteins - A complex of lipids and proteins, with greater amounts of lipid than protein, that transports cholesterol in the blood. High levels are associated with an increased risk of atherosclerosis and coronary heart disease. Researchers have linked LDL particle size to the subsequent development of heart disease.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 119 | 118
percent change | 1.5 [-0.5 to 4.1] | 0.5 [-1.0 to 2.0]

16. Secondary Outcome: Percent Change in Lipoprotein-Phosphoslipase A2 From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Lipoprotein Phosphoslipase A2 - modified form of LDL.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 119 | 118
percent change | -20.7 [-27.5 to -10.0] | -9.7 [-17.6 to -0.6]

17. Secondary Outcome: Percent Change in High Density Lipoprotein (HDL) Particle Concentration Total From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: High Density Lipoprotein partical size suggests the bigger the better. HDL is a complex of lipids and proteins in approximately equal amounts that functions as a transporter of cholesterol in the blood. High levels are associated with a decreased risk of atherosclerosis and coronary heart disease.
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 119 | 118
percent change | 1.0 [-8.9 to 8.4] | 5.1 [-1.3 to 11.9]

18. Secondary Outcome: Percent Change in High Density Lipoprotein (HDL) Particle Size From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Partical size suggests the bigger the better. HDL is a complex of lipids and proteins in approximately equal amounts that functions as a transporter of cholesterol in the blood. High levels are associated with a decreased risk of atherosclerosis and coronary heart disease.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 119 | 118
percent change | 0.0 [-1.2 to 2.4] | 1.2 [0.0 to 2.4]

19. Secondary Outcome: Percent Change in Very Low Density Lipoproteins and Chylomicron Particle Concentration Total From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Very low density lipoproteins are plasma lipoproteins with a high lipid content, associated with atherosclerosis. Chylomicrons are One of the microscopic particles of emulsified fat found in the blood and lymph and formed during the digestion of fats.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 119 | 118
percent change | -32.4 [-50.5 to -14.6] | -25.9 [-39.0 to -4.0]

20. Secondary Outcome: Percent Change in Very Low Density Lipoproteins Size From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Very low density lipoproteins are plasma lipoproteins with a high lipid content, associated with atherosclerosis.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 119 | 118
percent change | -17.5 [-26.0 to -9.5] | -3.3 [-11.5 to 10.1]

21. Secondary Outcome: Percent Change in Intermediate Density Lipoprotein Particle Concentration From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Intermediate Density Lipoprotein, or IDLs, transport cholesterol and triglycerides through the body. IDLs are a type of cholesterol that are a product of VLDL degradation and result in LDL cholesterol when broken down.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 114 | 112
percent change | -60.4 [-87.9 to -18.6] | -50.3 [-77.2 to -20.5]

22. Secondary Outcome: Percent Change in Remnant-like Particle Cholesterol From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Remnant-like particle cholesterol within the plasma has been identified as a cardiovascular risk factor.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 118 | 119
percent change | -50.0 [-61.1 to -38.5] | -38.9 [-53.1 to -18.5]

23. Secondary Outcome: Percent Change in Total Adiponectin From Baseline to Week 8 During 10 mg Atorvastatin Treatment Period
Description: Adiponectin is a protein hormone that modulates a number of metabolic processes, including glucose regulation and fatty acid catabolism.
Time Frame: Baseline and Week 8
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 119 | 118
percent change | -5.1 [-15.2 to 8.2] | -1.6 [-12.6 to 7.7]

24. Secondary Outcome: Percent Change in Non-High Density Lipoprotein Cholesterol From Baseline to Week 12 During 20 mg Atorvastatin Treatment Period
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 117 | 118
percent change | -46.9 [-52.2 to -40.1] | -39.0 [-45.3 to -33.5]

25. Secondary Outcome: Percent Change in Non-High Density Lipoprotein Cholesterol From Baseline to Week 16 During 40 mg Atorvastatin Treatment Period
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 113 | 112
percent change | -50.4 [-57.6 to -43.3] | -46.3 [-51.7 to -40.3]

ADVERSE EVENTS:
Arm/Group | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Serious Adverse Events (participants affected / at risk) | 4 | 2
Other Adverse Events (participants affected / at risk) | 0/123 | 0/122
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Lovaza(Omacor) + Atorvastatin | Placebo + Atorvastatin
Cholecystitis Acute (Hepatobiliary disorders) | 0/122 | 1/122
Syncope (Nervous system disorders) | 0/122 | 1/122
Peripheral Ischemia (Vascular disorders) | 1/122 | 0/122
Lobar Pneumonia (Infections and infestations) | 1/122 | 0/122
Chest Pain/ Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/122 | 0/122
Labyrinthitis (Infections and infestations) | 1/122 | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centres of a multi-centre trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.